CLINICAL TRIAL: NCT01831258
Title: Comparison Study of the ICON™ CPAP Series With and Without SensAwake™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FPH-SA13-01
Record Dates: First submitted 2013-04-02; First posted 2013-04-15 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- SensAwake On (Experimental): The comfort feature 'SensAwake' will be turned on
  Interventions: Device: SensAwake On
- SensAwake Off (Active Comparator): The comfort feature 'SensAwake' will be turned off
  Interventions: Device: SensAwake Off

INTERVENTIONS:
Device: SensAwake On
  Arms: SensAwake On
Device: SensAwake Off
  Arms: SensAwake Off

SUMMARY:
Conceptually, awareness of pressure occurs only during wakefulness. Thus reducing the pressure during wakefulness may improve therapy comfort and potentially adherence without compromizing therapy efficacy. SensAwake™ is a unique pressure relief technology developed by Fisher & Paykel Healthcare which detects irregularity in the flow signal indicative of the transition from sleep to wake. When the transition from sleep to wake is detected the device promptly reduces the pressure to help facilitate a return to sleep.

The purpose of this study is to compare adherence and sleep quality outcomes in patients treated by CPAP with and without SensAwake technology.

It is hypothesised that participants with SensAwake on will have improved adherence and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years with moderate-to-severe OSA (AHI equal to or greater than 10 per hour).
* Successful in-lab titration polysomnography (PSG)
* General (at home) sleep habits of:
* At least 7 hours in bed on most nights
* Lights out at 12 midnight or earlier
* Fluency in both written and spoken English.

Exclusion Criteria:

* Participants prescribed and fitted with any PAP device in the past 2 years
* Contraindicated for CPAP or AutoCPAP therapy.
* Any known factor or disease that might interfere with treatment adherence, study conduct or interpretation of the results such as severe psychiatric disease, history of non adherence to medical regimens, or unwillingness to comply with study requirements as determined by the principal investigator.
* Other significant sleep disorder(s) that would interfere with their ability to wear CPAP as determined by the principal investigator.
* Patients who are prescribed hypnotics and sedating medications.
* Any surgery of the mouth, nose, sinuses or airways (for OSA, snoring or otherwise) in the past 12 months.
* If participants are required, by the nature of their employment, to comply with therapy. For example truck drivers or airline pilots.
* If the physician objects to their patient taking part in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pulmonary Associates, Glendale, Arizona
  - SleepMed of Central Georgia, Macon, Georgia
  - Sleep Med of South Carolina, Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- SensAwake On, Then Followed by SensAwake Off: The comfort feature 'SensAwake' will be turned on, followed by it off.
- SensAwake Off, Then Followed by SensAwake On: The comfort feature 'SensAwake' will be turned off, then followed by on.
Period: Overall Study
Arm/Group | SensAwake On, Then Followed by SensAwake Off | SensAwake Off, Then Followed by SensAwake On
Started | 35 | 35
Completed | 30 | 32
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either SensAwake On or SensAwake Off
Arm/Group | All Study Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only collected 65 participants data on age
  years
    number analyzed (Participants) | 65
    (all) | 50.78 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only collected n=68. Missing data for 2 participants.
  Participants
    number analyzed (Participants) | 68
    Female | 22
    Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Adherence to CPAP Treatment
Description: Average used minutes (all days) taken from the CPAP device.
Time Frame: 2 weeks
Population: Adherence data could only be obtained for 61 participants
Measure: Mean (Standard Error); unit: mins
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 61 | 61
mins | 272.672 (17.055) | 289.087 (15.239)

2. Secondary Outcome: Daytime Sleepiness (Subjective Sleep Quality)
Description: Collected through the Epworth Sleepiness Scale (ESS) which is a subjective questionnaire and the participant answer 8 question with rating on the chance of dozing (from 0= no chance of dozing to 3 = high chance of dozing). The total is added with a range from 0-24. A total score of 0 means that the participant is not experiencing day time sleepiness, while total score of 24 means that the participant si extremely sleepy during the daytime.
Time Frame: 4 weeks
Population: Data for 65 participant were available
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 65 | 65
units on a scale | 6.9 (0.6) | 6.4 (0.6)

3. Secondary Outcome: Insomnia Severity Index (Subjective Sleep Quality)
Description: Collected through the Insomnia Severity Index (ISI). There are seven question with each question having a scale of 0 (no issue) to 4 (very severe). The total score is added up. If the participant has a total score of 0-7 = no clinical significant insomnia, total score of 8-14 = sub threshold insomnia, total score of 15-21 = clinical insomnia (moderate), total score of 22-28 = clinical insomnia (severe).
Time Frame: 4 weeks
Population: Data for 63 participant were available
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 63 | 63
units on a scale | 7.8 (0.8) | 7.3 (0.7)

4. Secondary Outcome: OSA Impact of Daily Life
Description: Collected through the Short Functional Outcomes of Sleep Questionnaire (FOSQ-10). The questionnaire has 10 questions which ask how daytime sleepiness has impacted their quality of life. Each question has a scale of 1 = yes extreme to 4 = No. Lower total score (min 10) means that the disease is affecting your quality of life while a higher total score (maximum 40) means that the disease is not affecting your quality of life.
Time Frame: 4 weeks
Population: Data for 62 participant were available
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 62 | 62
units on a scale | 32.7 (1.0) | 34.6 (0.9)

5. Secondary Outcome: OSA Impact of Daily Life (Fatigue)
Description: Collected through the Fatigue Severity Scale (FSS). There are 9 question on fatigue with each question having a scale of 1 = strongly disagree and 7 = strongly agree. A lower total score (minimum of 9) = low severity with fatigue while a higher total score (maximum of 63) indicates a higher severity with fatigue.
Time Frame: 4 weeks
Population: Data for 64 participant were available
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 64 | 64
units on a scale | 29.3 (1.6) | 28.2 (1.9)

6. Secondary Outcome: Subjective Treatment Efficacy - Patient Global Impression of Change (PGI) - Severity
Description: Collected through the Patient Global Impression of Change (PGI).The questions ask "Since beginning CPAP therapy, how would you describe the chance (if any) in symptoms related to your OSA. The questions has a scale of 1 = no change (or condition has got worse) to 7 = a great deal better and a considerable improvement that has made all the difference.
Time Frame: 4 weeks
Population: Data for 64 participant were available
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 64 | 64
units on a scale | 4.3 (0.2) | 4.4 (0.2)

7. Other Pre Specified Outcome: Leak
Description: The amount of Continuous Positive Airway Pressure (CPAP) leak was obtained through the device
Time Frame: One night
Population: Obtained only 61 participant CPAP data.
Measure: Mean (Standard Error); unit: L/min
Groups:
- SensAwake On: The comfort feature 'SensAwake' will be turned on
  SensAwake On
- SensAwake Off: The comfort feature 'SensAwake' will be turned off
  SensAwake Off
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 61 | 61
L/min | 41.72 (2.52) | 48.91 (3.01)

8. Other Pre Specified Outcome: Apnea Hypopnea Index (AHI)
Description: Collected through the device
Time Frame: 2 weeks
Population: Only 61 participant data was available.
Measure: Mean (Standard Error); unit: events/hour
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 61 | 61
events/hour | 5.182 (0.590) | 3.563 (0.464)

9. Post Hoc Outcome: Adherence in Patients With Signs of Moderate Clinical Insomnia
Description: Adherence from the device (during their first treatment arm) in patients with moderate clinical insomnia (Insomnia Severity Index 15 or over)
Time Frame: 4 weeks
Population: Only participant with moderate clinical insomnia (Insomnia Severity Index of 15 and over) were included in the post-hoc.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 18 | 12
minutes | 322.89 (26.46) | 282.25 (30.58)

10. Post Hoc Outcome: Adherence in Patients With Signs of Moderate Clinical Insomnia
Description: Adherence from the device (during their entire study period) in patients with moderate clinical insomnia (Insomnia Severity Index 15 or over)
Time Frame: 8 weeks
Population: Only participant with moderate clinical insomnia (Insomnia Severity Index of 15 and over) were included in the post-hoc.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 18 | 12
minutes | 304.787 (28.75) | 238.42 (35.57)

11. Secondary Outcome: Subjective Treatment Efficacy - Patient Global Impression of Change (PGI) - Change
Description: Collected through the Patient Global Impression of Change (PGI).The questions ask "Since beginning CPAP therapy, how would you describe the change (if any) in overall quality of life related to your OSA?". The questions has a scale of 1 = no change (or condition has got worse) to 7 = a great deal better and a considerable improvement that has made all the difference.
Time Frame: 4 weeks
Population: Data for 64 participant were available
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SensAwake On | SensAwake Off
Number analyzed (Participants) | 64 | 64
units on a scale | 4.2 (0.2) | 4.3 (0.2)

ADVERSE EVENTS:
Time Frame: 1 year and 1 month
Arm/Group | SensAwake On | SensAwake Off
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/70
Other Adverse Events (participants affected / at risk) | 11/70 | 16/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SensAwake On (N=70) | SensAwake Off (N=70)
High Blood Pressure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Participant was hospitalized with symptoms of extremely high blood pressure. No formal diagnosis was given prior to discharge however subjects were placed on hypertension medication. PI deemed as not related to the device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SensAwake On (N=70) | SensAwake Off (N=70)
Mask related issues (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) — 11 events were related to the mask, it was not related to the device. There were sore on nose, skin breakdown from mask and mask irritations
Cold or Upper Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) — Cold or Upper Respiratory Infections. They were not related to the device
Broken Arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Broken Arm not related to the device
Dizziness upon Arousal (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Not related to the device
Pressure related problems (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — Feeling higher pressure from the device
Scheduled Achilles Tendon Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not related to the device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No